CLINICAL TRIAL: NCT03083964
Title: APP-ME: Addressing Place and People MicroEnvironments in Weight Loss Disparities
Brief Title: Addressing Place and People Micro Environments in Weight Loss Disparities
Acronym: APP-ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, NiCole Keith, Professor, Department of Kinesiology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1512254890
Record Dates: First submitted 2017-02-14; First posted 2017-03-20 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Obese
Keywords: Middle aged women; 35-64yrs; BMI= >30
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The participants are randomized to one of two treatment arms, usual care or intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcome assessor is blind to study assignment and investigators do not have access to randomization records.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Usual care involves a lifestyle coaching intervention delivered in primary care sites.
  Interventions: Behavioral: Usual Care
- Priming (Experimental): Priming involves usual care plus just in time reminder messages related to mindful eating and physical activity.
  Interventions: Behavioral: Priming

INTERVENTIONS:
Behavioral: Usual Care — Usual care is not considered an intervention. This arm of the study involves a lifestyle coaching intervention delivered in primary care sites to the subjects.
  Arms: Usual Care
Behavioral: Priming — The intervention is a just in time eating or physical activity reminder. Each individual participant reports physical activity goals as well as times that they most often eat. This information is used to select for that individual the best time to send an eating or physical activity reminder. The reminders come to the participant's smartphone or a study provided smartphone. Participants will receive reminder 2 to 4 times per day depending on their goals and behavior pattern.
  Arms: Priming

SUMMARY:
The purpose of this study is to A) capture obesogenic cues that occur in daily life, and B) to deliver cue alerts. Investigators hypothesized that A) black women experience more cues, B) racial disparities in obesity are reduced in models that adjust for cues, and C) the priming arm will achieve a weight loss of 2kg or more. Investigators will explore whether racial disparities in weight loss differ between the groups receiving usual care or those receiving cues.

DETAILED DESCRIPTION:
Aim 1: After participants have been consented over the phone or in clinic, the Research Assistants (RA) will schedule a baseline assessment. Baseline interviewer administered survey questions, assessments, and equipment set-up will be completed in participants' homes to allow a physical environment assessment of the home. Assessments and surveys will be carried out using Research Electronic Data Capture (REDCap; see Resources). The in-home baseline assessment piloted for the proposed study takes 1 to 1.5 hours. Global Positioning System (GPS) locating, accelerometry, bite monitoring, and EMA surveys will operate through the mHealth app over the immediate 2-4 week period. For GPS locating, the mHealth app uses software that identifies and sends the longitude and latitude at the time of EMA response to a secure IU server. Software then determines the address of the location and whether it is the participant's home, work, restaurant, retail store, etc. For messaging, the mHealth app uses "Push Notification" to deliver EMA requests to the device (i.e., smartphone). This bypasses the phone carrier's Short Message Service (SMS) gateway, which is not always reliable or secure. The mHealth app makes sure the messages are delivered and secure. Participants receive a notification and open the application to answer the EMA questions. The database is located in a secure network within Indiana University servers. None of the data are stored inside the smartphone at rest. The actual questions are very brief with radio button responses.

At the end of the 2-4 week window, RAs will return to the home to collect the accelerometer and bite counter which takes about 1 hour. The accelerometer and bite counter are to be marked by the RA with the study participants ID and data are retrieved. At this time, participants who responded to 75% or more of the messages over the 2-4 week period, will be randomized to Usual Care (UC) or Priming Arm for Aim 2 and given instruction on the next steps of study participation. Randomization will be carried out within each race group to ensure a balance in the number of subjects between the two treatment arms. The Investigator will computer-generate randomization lists in field envelopes to be provided to the RAs for treatment assignment.

Aim 2: The second aim of the study will last 6 months. Both UC and Priming arms will have full access to Healthy-Me coaches and classes as well as receive training and access to the mHealth app. When study participation is excluded, all apps and associated data will be removed from the smartphone. At no time will Patient Health Information (PHI) be stored on the smartphone. Smartphones will only be identified by study ID number and the developer will only have access to the participants' study ID number and smartphone data collected by the mHealth app. Subjects in UC and Priming will undergo similar assessments and procedures; however, the Priming arm participants will, in addition receive 6-8 message alerts per day. The application and notifications that will be used in the Priming arm will be built from each participants own library to be delivered at times and in locations that their Aim 1 data indicate they often experience an eating or sedentary cue. In short, this intervention counters an obesogenic cue with a "healthy" prime in real-time and location.

Finally, following 6 months of UC or Priming, blinded RAs will return to participants home to complete 6-month follow-up assessment and collect all study related equipment. The final assessment and surveys will take about 1-1.5 hours and all data captured will also be carried out in REDCap.

ELIGIBILITY:
Inclusion Criteria:

* Electronic Screener Data (EMR):

  1. Aged 35 to 64 years.
  2. Female.
  3. BMI ≥ 30.
  4. Healthy-Me referral or Eligible for Healthy-Me

     Self-reported Screener Data:
  5. English as primary language.
  6. Self-identified non-Hispanic black or African-American, or non-Hispanic white.
  7. A permanent address.

Exclusion Criteria:

* Electronic Screener Data (EMR):

  1. Severe illness that might be associated with weight loss, such as cancer.
  2. Use of weight loss medications (rare due to cost of the medications).
  3. History of bipolar disorder or psychosis.

     Self-reported Screener Data:
  4. Severe cognitive impairment (≥3 errors on a 6-item cognitive screen).
  5. Unwilling or unable to provide informed consent.
  6. Bariatric surgery already completed or planned within 12 months.
  7. Pregnant or nursing in past 6 months, or plans to become so within 12 months.
  8. Residence outside of Marion County, Indiana.
  9. Substance abuse (for alcohol; ≥2 on CAGE questionnaire).
  10. Current smoking or tobacco use.

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Enrolling females to capture obesogenic cues as they occur in daily life among 150 obese black and 150 obese white women ages 35-64 years who have received an FQHC provider referral to the Healthy Me weight management program.
Enrollment: 350 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Proportion of participants that lose 2 kilograms of weight between baseline and 6 month follow-up | baseline and 6 months
  Participants are weighed at baseline and 6 months to access if proportion is losing 2kg of body weight or more by 6 months.

SECONDARY OUTCOMES:
Physical activity frequency | 6 months
  Outcomes include ecological momentary assessments that query up to 12 times per day to address physical activity using smartphones.
Eating Frequency | 6months
  Participants will self-report eating behavior for 3 week periods at baseline and follow-up at 6 month.
Depression | 6 months
  Depression is measured using the patient health questionnaire PHQ-4
Anxiety | 6 months
  Anxiety is measured using the patient health questionnaire PHQ-4

CONTACTS AND LOCATIONS:
Locations (1):
- Daniel Clark, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clark DO, Keith NR, Ofner S, Hackett J, Li R, Agarwal N, Tu W. Environments and situations as correlates of eating and drinking among women living with obesity and urban poverty. Obes Sci Pract. 2021 Sep 1;8(2):153-163. doi: 10.1002/osp4.557. eCollection 2022 Apr. PMID 35388340
- [Derived] Srinivas P, Bodke K, Ofner S, Keith NR, Tu W, Clark DO. Context-Sensitive Ecological Momentary Assessment: Application of User-Centered Design for Improving User Satisfaction and Engagement During Self-Report. JMIR Mhealth Uhealth. 2019 Apr 3;7(4):e10894. doi: 10.2196/10894. PMID 30942698